CLINICAL TRIAL: NCT05733429
Title: Eye-Cervical Re-education Versus Motor Imagery Therapy on Pain, Function, and Proprioception in Chronic Mechanical Neck Pain: A Randomized Controlled Trial
Brief Title: Eye-Cervical Re-education Versus Motor Imagery Therapy on Proprioception in Chronic Mechanical Neck Pain
Acronym: MNP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, Nabil mahmoud ismail, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004164
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
Keywords: Eye-Cervical Re-education; Motor Imagery Therapy; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: eye cervical re-education and motor imagery therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eye cervical re-education (Experimental): patients will receive eye cervical re-education three times a week for four weeks
  Interventions: Other: eye cervical re-education; Other: conventional physical therapy
- motor imagery therapy (Experimental): patients will receive motor imagery therapy three times a week for four weeks
  Interventions: Other: motor imagery therapy; Other: conventional physical therapy
- conventional physical therapy (Active Comparator): patients will receive conventional physical therapy three times a week for four weeks
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: eye cervical re-education — patients will receive eye-cervical re-education in the form of 10 exercises at three phases; the first phase will include stimulation of ocular mobility, the second phase will consist of Cervical mobility exercise with restricted eye movement and the third phase will include stimulation of eye and neck movement co-ordination
  Arms: eye cervical re-education
Other: motor imagery therapy — the patients will receive motor imagery therapy for four weeks; the first week will receive kinesthetic imagery, the second week will receive visual imagery, the third week will receive action observation exercises with motor imagery and the fourth week will receive motor control exercises in front of a mirror.
  Arms: motor imagery therapy
Other: conventional physical therapy — the patients will receive conventional physical therapy programs in the form of hot packs, therapeutic massage, cervical isometric strengthening exercises, and scapular stabilization exercises.

SUMMARY:
this study will be conducted to investigate the effect of eye-cervical re-education versus motor imagery therapy on pain intensity level, pain pressure threshold, neck disability, cervical proprioception, and scapular protraction in patients with chronic mechanical neck pain.

DETAILED DESCRIPTION:
Chronic neck pain is a common problem in modern and industrialized countries and among employed individuals. Pain is classified as chronic neck pain persists for more than 3 month, it may be felt all the time or worsen with certain activities. The cervical spine has an important role in providing the proprioceptive input and this is reflected in the abundance of cervical mechanoreceptors and their central and reflex connections to the vestibular, visual, and central nervous systems. Eye-cervical re-education program (ECRP) refer to a therapeutic procedure for correcting posture cephalic level in patients with cervical pain by improving eye-neck proprioception that reduced symptoms experienced by patients and improvement of the quality of cervical afferent input into the central nervous system. Motor imagery is the mental realization of motion without any motion occurs. It has two categories: kinesthetics and visual imagery. Kinaesthetic imagery is the situation of feeling a motion. Visual imagery has two types: internal visual and external visual. In the internal visual imagery, the motion is visualized within the body by seeing feet and arms. The external visual imagery is that one sees himself/herself from outside. one hundred and twenty patients will be allocated randomly into three groups; group A will receive eye cervical re-education and conventional therapy, group B will receive motor imagery therapy and conventional therapy and group C will receive conventional therapy only three times a week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age will range from 18 to 70 years
2. Patients of both sexes.
3. Neck pain diagnosed by physician greater than 3 months in duration.
4. Active or latent myofascial trigger points (MTrPs) in at least one of the following muscles: upper trapezius, levator scapulae, or splenius capitis. Both active and latent MTrPs were considered because latent MTrPs have been associated with the development of sensory motor dysfunction and may contribute to different chronic musculoskeletal pain disorders

Exclusion Criteria:

1. Dizziness syndrome.
2. Post-traumatic as whiplash
3. Neurological, infectious, or tumor cervical pain.
4. Pregnant women.
5. Patients having speech and understanding problems.
6. Past history of neck surgery
7. Dizziness syndrome.
8. Post-traumatic as whiplash.
9. Neurological, infectious, or tumor cervical pain.
10. Pregnant women.
11. Patients having speech and understanding problems.
12. Past history of neck surgery .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-02 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
joint position error | up to four weeks
  The Cervical Joint Position Error (JPE) Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability. Cervicocephalic proprioception describes one's sense of position of their head and neck in space. The Cervical JPE Test measures the ability of a blindfolded patient to accurately relocate their head position back to a predetermined neutral point after cervical joint movement. The test is most commonly performed with head movement in the transverse and sagittal planes by cervical range of motion device (CROM).

SECONDARY OUTCOMES:
disability | up to four weeks
  The neck disability index (NDI) will be used for measuring neck disability and it is a self-patient-completed questionnaire that measures patients' functional status. It contains 10 questions regarding pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each question has six answer choices scored from 0 to 5 as 0 indicates no disability and 5 indicates complete disability. All sections are scored then totaled on a scale from 0 to 50, as zero is the best possible score and 50 is the worst one
pain intensity | up to four weeks
  Visual Analogue Scale which is a 100-mm horizontal line will be used for measuring pain intensity. The patients will be instructed to represent their pain intensity level by marking anywhere on the line with "no pain" on the left side and "worst pain" on the right side
rounded shoulder | up to four weeks
  tape measurement will be used to to assess rounded shoulder: Subjects will be requested to stand normally with their hands hanging beside their bodies to test for rounded shoulder posture. Then, sternal notch, coracoid process, posteriolateral angle of the acromion process and the adjacent thoracic spinous process will be palpated and marked. The distance between sternal notch and coracoid process, and the distance between the posterolateral angle of the acromion process and the adjacent thoracic spinous process will measured by using tape
pressure pain threshold | up to four weeks
  pressure algometer device will be used for measuring pressure pain threshold